CLINICAL TRIAL: NCT01783041
Title: A Double-Blind, Controlled, Randomized Clinical Trial of the Effect of Early L-Carnitine Supplementation on Neurodevelopmental Outcomes in Very Preterm Infants
Brief Title: Effect of Early L-Carnitine Supplementation on Neurodevelopmental Outcomes in Very Preterm Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-07-234
Record Dates: First submitted 2013-01-25; First posted 2013-02-04 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Prematurity; Neurodevelopmental Disorder; Carnitine Deficiency
Keywords: Prematurity; Carnitine supplementation; Neonatal Intensive Care; MRI; Amplitude-integrated EEG; NICU Network Neurobehavioral Scale; Bayley Scale of Infant Development III
MeSH Terms: conditions — Premature Birth; Neurodevelopmental Disorders; Systemic carnitine deficiency | interventions — Carnitine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- 5% dextrose (Placebo Comparator): Infants randomized to the placebo group will receive 5% dextrose intravenously. If infant is receiving 100 cc/kg/day of enteral feeds before the supplementation endpoint, an equivalent volume of placebo (5% Dextrose) will be given to the study patients.
  Interventions: Drug: 5% Dextrose
- L-carnitine (Experimental): Infants randomized to the study group will receive L-carnitine intravenously. If infant is receiving 100 cc/kg/day of enteral feeds before the supplementation endpoint, an equivalent dose of enteral L-carnitine will be given to the study patients.
  Interventions: Drug: L-carnitine

INTERVENTIONS:
Drug: L-carnitine — Infants will receive L-carnitine 50 micromoles/kg/day, divided into three doses, intravenously for a minimum of 2 weeks or until they achieve enteral feeding volume of 100 cc/kg/day. If infant is receiving 100 cc/kg/day of enteral feeds before the supplementation endpoint, an equivalent dose of enteral L-carnitine will be given to the study patients.
  Other Names: Levocarnitine; Carnitor
  Arms: L-carnitine
Drug: 5% Dextrose — Infants will receive 5% dextrose (placebo) three times a day (volume equivalent to the experimental drug) intravenously for a minimum of 2 weeks or until they achieve enteral feeding volume of 100 cc/kg/day. If infant is receiving 100 cc/kg/day of enteral feeds before the supplementation endpoint, an equivalent volume of enteral placebo (5% Dextrose) will be given to the study patients.
  Arms: 5% dextrose

SUMMARY:
Preterm infants are vulnerable to brain injury, nutritional deficiencies and poor early growth which places them at increased risk for developmental problems later in life. The micronutrient carnitine, which is present in breast milk and stored in the fetus late in pregnancy, has been shown to protect against brain injury in animal studies. Without supplementation, almost all preterm infants develop carnitine deficiency soon after birth. Thus it is important to determine if carnitine supplementation protects against brain injury and improves developmental outcomes in these vulnerable preterm infants. We hypothesize that preterm infants supplemented early with L-carnitine while receiving parenteral nutrition will not develop carnitine deficiency and will have improved growth in the first two weeks of life and higher scores on developmental tests when compared to control infants who did not receive carnitine.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that preterm infants supplemented with early physiologic doses of L-carnitine while on parenteral nutrition will have improved short-term growth parameters and significantly higher neurobehavioral scores when compared with control infants.

Methods/Design: This is a prospective, randomized controlled clinical trial involving infants with gestational age (GA) <32 wks who are born at either the Jack D. Weiler Hospital or the Wakefield Division of Montefiore and admitted to theirNeonatal Intensive Care Unit. Informed consent will be obtained from the parents of eligible patients as early as possible within 72 hours of birth. Infants whose parents have signed an informed consent form will be randomized to receive either carnitine supplementation (50 μmol/kg/day) versus placebo within 72-96 hours of birth.

Randomization: As previously described by Pande et al., enrolled patients will be randomized to either the treatment group (L-carnitine, 50 μmol/kg/day) or placebo group (5% glucose, similar volume as the L-carnitine group).28 Patients who meet study entry criteria and have signed informed parental/guardian consent will be enrolled in the study. Because gestational age and small for gestational age (SGA) status will impact our outcome measures, we will ensure they are equally distributed in the arms of the study by stratifying based upon these variables. We will analyze the two study arms using an intent-to-treat analysis. Therefore, enrolled patients will be stratified into fourgroups: gestational age 23 to 26 6/7 weeks, gestational age 27 to 29 6/7weeks, gestational age 30 to 31 6/7 weeks and small for gestational age (SGA). Patients within each stratum will be randomized by the pharmacist using a computerized block-generation with sets of 4. In the case of multiple births, all infants must meet study criteria, and the infants will be randomized as a set. One infant of the multiple-birth set will be randomly chosen for inclusion in the analysis. A recruitment log of all screened infants will be maintained. Clinicians and the nursing staff will be unaware of the arm of the treatment protocol to which the patient is assigned. Codes will be unblinded only after all patients have reached the study end-point, or at the request of the Data Safety Monitoring Board.

Study supplementation: Infants randomized to the treatment group will receive 50 μmol/kg/day of L-carnitine intravenously for 2 weeks, and infants randomized to placebo will received 5% glucose, similar volume to the L-carnitine group. At two weeks, sufficient carnitine is provided in enteral feeds of either breast milk or infant formula. If no intravenous access is available before the supplementation endpoint, the equivalent dose of enteral study supplement (L-carnitine or placebo) will be administered.41 Parenteral and enteral nutrition will be provided according to standard NICU protocol.

Of note, as many as 10% of the infants in the study will likely continue to rely primarily on parenteral nutrition beyond the proposed two-week supplementation period. Enteral feeds may be withheld from these infants due to underlying illnesses such as sepsis or gastrointestinal disorders like necrotizing enterocolitis. Due to the presence of underlying illness, these infants are at an even higher risk for developing developmental delays. Therefore, in study patients who are not receiving adequate enteral nutrition (100 cc/kg/day of enteral intake) after 2-weeks of study supplements, carnitine supplementation will be continued until these infant are receiving adequate enteral feeds; at this point, their physiologic carnitine requirements will be met by enteral nutrition alone.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at equal to or less than 30 weeks gestation and with birth weight < 1250 grams
* Less than 72 hours of age
* Signed parental consent

Exclusion Criteria:

* Critically ill infants with life expectancy less than 72 hours
* Inability to obtain consent within 72 hours of birth
* Potentially life-threatening congenital anomalies
* Known hereditary metabolic disorders
* Known chromosomal abnormalities
* Terratogen exposure with symptomatic substance withdrawal
* Congenital viral infections
* Microcephaly
* Grade IV intraventricular hemorrhage or seizures documented within the first 72 hours of life

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2013-01; Primary Completion 2020-12 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Fuloria, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Montefiore Medical Center - Jack D. Weiler Division, The Bronx, New York
  - Montefiore Medical Center - Wakefield Division, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants born at <32 weeks gestation admitted to the Neonatal Intensive Care Unit (NICU) at Weiler and Wakefield Divisions of Montefiore Medical Center were enrolled in this study.
Period: First 2 Weeks of Life
Arm/Group | 5% Dextrose | L-carnitine
Started | 72 | 72
Completed | 69 | 71
Not Completed | 3 | 1
Period: NNNS Examination at Term Equivalent Age
Arm/Group | 5% Dextrose | L-carnitine
Started | 69 | 71
Completed | 60 | 59
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5% Dextrose | L-carnitine | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72 | 72 | 144
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 36 | 38 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 37 | 72
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 28 | 58
  White | 38 | 40 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 72 | 72 | 144

OUTCOME MEASURES:

1. Primary Outcome: Time to Regain Birthweight in Infants Who Receive L-carnitine Supplementation Compared to Controls
Description: Time (in days) for infants in both arms of the study to regain birthweight - data presented as mean +/- SD.
Time Frame: up to 3 weeks of age
Population: The discrepancy in the number of infants enrolled in each arm of the study and the number with data for this outcome is because of early deaths in the study as well as some parents withdrawing consent from the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 5% Dextrose | L-carnitine
Number analyzed (Participants) | 68 | 68
days | 8.12 (3.5) | 8.4 (3.3)
Statistical Analysis 1: Comparison: 5% Dextrose vs L-carnitine; Test type: Other; p < 0.05, ANOVA — These are calculated p values; Differences in continuous and categorical variables were compared using ANOVA and either Chi square test or Fisher's exact test, respectively

2. Primary Outcome: Neurodevelopment Indices in Infants Who Receive L-carnitine Supplementation Compared to Controls (NNNS)
Description: NICU Network Neurobehavioral Scale (NNNS) was administered to study participants at term equivalent age (38 weeks +/-1 week corrected age). The NNNS is a 128-item standardized assessment to evaluate the neurobehavioral status of healthy and high-risk infants. Summary scores include: Attention (range 2.25-8; higher score better), Arousal (range 2-5; lower score better), Regulation (range 3.31-6.92; higher score better), Handling (range 0-0.88; lower score better), Quality of movement (range 3-6; higher score better), Excitability (range 0-9; lower score better), Lethargy (range 0-12; lower score better), Nonoptimal reflexes (range 0-10; lower score better), Asymmetric reflexes (range 0-6; lower score better), Hypertonicity (range 0-2; lower score better), Hypotonicity (range 0-3; lower score better), and Stress/abstinence scale (range 0-0.22; lower score better).
Time Frame: at term equivalent age (38 weeks +/-1 week corrected age)
Population: The discrepancy in the numbers analyzed for this outcome compared to the enrolled participants in each study arm is related to: (1) mortality, (2) parents revoking consent, and (3) some patients were too sick for this evaluation to be performed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5% Dextrose | L-carnitine
Number analyzed (Participants) | 60 | 59
score on a scale
  Attention | 4.66 (1.62) | 4.29 (1.41)
  Stress abstinence | 0.073 (0.074) | 0.079 (0.064)
  Quality of Movement | 4.6 (0.63) | 4.6 (0.64)
  Arousal | 3.95 (0.6) | 3.93 (0.61)
  Regulation | 5.5 (0.77) | 5.5 (0.84)
  Handling | 0.35 (0.28) | 0.36 (0.23)
  Hypertonicity | 0.12 (0.32) | 0.14 (0.43)
  Hypotonicity | 0.57 (0.87) | 0.22 (0.46)
  Asymmetrical Reflexes | 0.35 (0.79) | 0.37 (0.72)
  Non-Optimal Reflexes | 3.95 (2.25) | 4.2 (2.2)
  Excitability | 2.6 (2) | 2.59 (1.99)
  Lethargy | 4.8 (3) | 5.2 (2.6)
Statistical Analysis 1: Comparison: 5% Dextrose vs L-carnitine; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney) — These are calculated p values; This analysis applies to all sub-scales that were compared between the 2 study groups

3. Secondary Outcome: Brain Volumes in Infants Who Received L-carnitine Supplementation Compared to Controls
Description: Brain MRI findings including brain volumes of the cerebellum, thalamus and basal ganglia were compared in infants who received L-carnitine supplementation compared to controls.
Time Frame: at corrected age (38 weeks +/- 1 week)
Population: Not all enrolled subjects had brain MRIs performed - 63 infants in both study arms had brain MRIs where brain volumes could be calculated.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | 5% Dextrose | L-carnitine
Number analyzed (Participants) | 63 | 63
milliliters
  Cerebellar volume | 19372 (5806) | 18189 (3826)
  Thalamus volume | 6050 (1139) | 5832 (897)
  Basal ganglia volume | 8611 (1460) | 8217 (1192)
Statistical Analysis 1: Comparison: 5% Dextrose vs L-carnitine; Test type: Other; p < 0.05, t-test, 2 sided — Reported p values have been calculated; Differences between the groups were analyzed using a two sided t-test

4. Secondary Outcome: Rate of Head Growth in Infants Who Receive L-carnitine Supplementation Compared to Controls
Description: Head circumference was measured at 36 weeks corrected age in both study groups (L-carnitine vs. placebo).
Time Frame: 36 weeks corrected age
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | 5% Dextrose | L-carnitine
Number analyzed (Participants) | 68 | 68
centimeters | 30.6 (1.68) | 30.4 (1.76)
Statistical Analysis 1: Comparison: 5% Dextrose vs L-carnitine; Test type: Other; p < 0.05, ANOVA — These are calculated p values; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Until hospital discharge, generally upto approximately 44 weeks post-menstrual age.
Arm/Group | 5% Dextrose | L-carnitine
All-Cause Mortality (participants affected / at risk) | 3/72 | 1/72
Serious Adverse Events (participants affected / at risk) | 18/72 | 24/72
Other Adverse Events (participants affected / at risk) | 4/72 | 9/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5% Dextrose (N=72) | L-carnitine (N=72)
Bronchopulmonary Dysplasia (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 23 (23) — Moderate to severe bronchopulmonary dysplasia
Patent ductus arteriosus (Cardiac disorders) | 18 (18) | 24 (24) — Presence of moderate to large PDA
Intraventricular hemorrhage (Nervous system disorders) | 3 (3) | 3 (3) — Grade 3 or 4 IVH
Surgical necrotizing entercolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — NEC requiring surgical intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5% Dextrose (N=72) | L-carnitine (N=72)
Blood culture positive sepsis (Infections and infestations) | 4 (4) | 9 (9) — Blood culture positive sepsis

LIMITATIONS AND CAVEATS:
This is a single center study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT01783041/Prot_SAP_000.pdf